CLINICAL TRIAL: NCT05109195
Title: A Prospective, Observational Standard of Care Study of Patients With Major Depressive Disorder Who Have Had an Inadequate Response to a Selective Serotonin Reuptake /Serotonin-Norepinephrine Reuptake Inhibitor Antidepressant as a Control Arm for the Safety Assessments in the Seltorexant Phase 3 Program
Brief Title: A Standard of Care Study of Patients With Major Depressive Disorder Who Have Had an Inadequate Response to a Selective Serotonin Reuptake/Serotonin-Norepinephrine Reuptake Inhibitor Antidepressant
Status: Terminated | Type: Observational
Why Stopped: due to business reasons.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109066; 42847922MDD3009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- MDD Participants with Insufficient Response to SSRI/SNRI (antidepressant): Major Depressive Disorder (MDD) participants with insufficient response to a selective serotonin reuptake inhibitor (SSRI)/serotonin-norepinephrine reuptake inhibitor (SNRI) (antidepressant) and starting an adjunctive therapy will be observed to create an external control arm (ECA) based on real world data (RWD) from electronic health records (EHR) data during routine medical care (standard of care [SOC]) combined with scheduled research assessments.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Other: Standard of Care (SOC) — Participants will not receive any intervention as a part of this study. Participants will receive SOC treatment.

SUMMARY:
The purpose of this study is to assess the safety (adverse events, serious adverse events, deaths, suicidality) of participants with major depressive disorder (MDD) treated according to the standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of Major Depressive Disorder (MDD) without psychotic features as confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Treatment with an selective serotonin reuptake inhibitor (SSRI)/serotonin-norepinephrine reuptake inhibitor (SNRI) for at least 6 weeks at an adequate dose (per Massachusetts General Hospital-Antidepressant Treatment Response Questionnaire [MGH-ATRQ]). Specifically, one of the following in any formulation is allowed: SSRIs: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline; SNRIs: venlafaxine, desvenlafaxine, vilazodone, or vortioxetine
* In the opinion of the treating clinician, the participant requires augmentation of the current antidepressant treatment and plans to initiate augmentation treatment in the near future. The participant has agreed to receive augmentation treatment
* Is currently an outpatient receiving psychiatric care (not inpatient care settings)
* Has a body mass index (BMI) of 18-40 kilograms per meter square (Kg/m^2), inclusive

Exclusion Criteria:

* Taking more than one antidepressant (regardless of class) at therapeutic doses (therapeutic doses per MGH-ATRQ). A second antidepressant is allowed to be taken at a lower dose if for sleep or pain management
* Is currently taking a benzodiazepine at higher doses than the equivalent of 3 milligrams (mg) of lorazepam
* Current diagnosis of a psychotic disorder including MDD with psychosis, bipolar disorder, intellectual disability, dementia, autism spectrum disorder, borderline personality disorder, or somatoform disorders
* Has treatment resistant depression (TRD) as defined by lack of response (less than [<] 25 percent [%] improvement) of 2 or more antidepressants of adequate dose (per MGH-ATRQ) and duration (6 weeks) in this episode
* Current diagnosis of PTSD, obsessive compulsive disorder, fibromyalgia, anorexia nervosa, or bulimia nervosa. Participants may be enrolled if they have been in remission for the past year

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consists of participants who will have one of the augmenting agents started.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Spontaneously Reported Adverse Events (AEs) | Up to 1 year
  Number of participants with spontaneously reported AEs will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs Collected through Generic Assessment of Side Effects (GASE) | Up to 1 year
  Number of participants with AEs collected through GASE will be reported. The GASE is an instrument to assess side effects in clinical studies that allows the detection of drug induced AEs.
Number of Participants with Hospitalization for Psychiatric Reasons | Up to 1 year
  Number of participants with hospitalizations for psychiatric reasons will be reported.
Number of Participants with Hospitalization for Medical Reasons | Up to 1 year
  Number of participants with hospitalizations for medical reasons will be reported.
Number of Participants with Other Serious Adverse Events (SAEs) | Up to 1 year
  SAE is any untoward medical occurrence that at any dose results in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Number of Participants with Deaths | Up to 1 year
  Number of participants with deaths will be reported.
Number of Participants with Suicide Attempts and Completed Suicides | Up to 1 year
  Number of participants with suicide attempts and completed suicides will be reported.
Suicidality Assessment Using the Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to 1 year
  Suicidality assessment using the C-SSRS will be reported. C-SSRS is semi structured clinician-administered questionnaire designed to solicit the occurrence, severity, and frequency of suicide-related ideation and behaviors. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Worsening of suicidal ideation will be an increase in severity of suicidal ideation from baseline.
Number of Participants with Suicidal Ideation as Assessed by C-SSRS | Up to 1 year
  Number of participants with suicidal ideation as assessed by C-SSRS, particularly codes of 4 or 5 will be reported. C-SSRS is semi structured clinician-administered questionnaire designed to solicit the occurrence, severity, and frequency of suicide-related ideation and behaviors. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Worsening of suicidal ideation will be an increase in severity of suicidal ideation from baseline.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events of Special Interest (AESI) | Up to 1 year
  Number of participants with AESI: Cataplexy, Sleep paralysis, Complex sleep-related behaviors, Falls, Motor vehicle accidents will be reported.
Change from Baseline in Weight Over Time | Baseline (Week 1) up to 1 year
  Change from baseline in weight over time will be reported.
Percentage of Participants with Clinically Meaningful Change in Weight | Baseline (Week 1) to end of study (up to 1 Year)
  Percentage of participants with clinically meaningful change in weight (greater than or equal to [>=] 7 percent [%]) from baseline to end of study will be reported.
Change from Baseline in Hemoglobin Level Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in hemoglobin level over time will be reported.
Change from Baseline in Platelet and White Blood Cell (WBC) Count Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in platelet and WBC count with differential over time will be reported.
Change from Baseline in Hematocrit Level Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in hematocrit level over time will be reported.
Change from Baseline in Red Blood Cell (RBC) Count Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in RBC count over time will be reported.
Change from Baseline in Sodium, Potassium, Chloride and Bicarbonate Level Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in sodium, potassium, chloride and bicarbonate level over time will be reported.
Change from Baseline in Blood Urea Nitrogen (BUN), Creatinine, Glucose, Total and Direct Bilirubin, Calcium and Phosphate Level Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in BUN, creatinine, glucose, total and direct bilirubin, calcium and phosphate level over time will be reported.
Change from Baseline in Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase Level Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in AST, ALT, alkaline phosphatase level over time will be reported.
Change from Baseline in Albumin and Total Protein Level Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in albumin and total protein level over time will be reported.
Change from Baseline in Total Cholesterol, Low-density Lipoprotein Cholesterol, Triglycerides, High-density Lipoprotein Cholesterol Level Over Time | Baseline (Week 1), Week 26 and Week 52
  Change from baseline in total cholesterol, low-density lipoprotein cholesterol (calculated), triglycerides, high-density lipoprotein cholesterol level over time will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Brigham And Women's Hospital, Boston, Massachusetts
  - The University of Pittsburgh of the Commonwealth System of Higher Education, Pittsburgh, Pennsylvania
- Warneford Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No